CLINICAL TRIAL: NCT01098695
Title: Early Family-Centered Prevention of Drug Use Risk
Brief Title: Early Family-Centered Prevention of Drug Use Risk (Aka Early Steps)
Acronym: Early Steps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: University of Pittsburgh (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3R01DA016110 (NIH)
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Substance Use; Conduct Disorder; Depression; Anxiety
Keywords: parenting interventions; Family Check-Up; Early Intervention; Self-Regulation
MeSH Terms: conditions — Substance-Related Disorders; Conduct Disorder; Depression; Anxiety Disorders; Self-Control | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EcoFIT offered (Experimental)
  Interventions: Other: Ecological Family Intervention and Treatment (EcoFIT)
- No Feedback or services offered (No Intervention)

INTERVENTIONS:
Other: Ecological Family Intervention and Treatment (EcoFIT) — Includes the Family Check-Up (in-person intake, family video observations and Assessment questionnaires used to provide and tailored feedback using motivational interviewing techniques) as well as continued tailored intervention services using the Everyday Parenting Curriculum.
  Other Names: Family Check-Up (FCU)
  Arms: EcoFIT offered

SUMMARY:
The investigators are testing the efficacy of a family-based preventive intervention, which began when the children were age 2, with children at risk for developing significant conduct problems. Families who were originally recruited from Women, Infants and Children (WIC) were randomly assigned to a family-centered intervention developed by Dishion and colleagues (Dishion & Kavanagh, 2003; Dishion & Stormshak, 2006) referred to as an 'ecological approach to family intervention and treatment' (EcoFIT). The current study expands the Early Steps intervention into the elementary school years beyond what is currently available for a WIC service delivery venue, in which children are no longer eligible for services at age 6.

The investigators are testing the hypothesis that periodic, tailored, and adaptive interventions delivered to caregivers at school entry will (a) reduce the probability of elevated risk associated with early-onset problem behavior, including the eventual use of drugs and other health-risking behaviors; (b) reduce the likelihood of mental health problems such as childhood depression, anxiety, conduct problems and co-morbidity; and (c) promote children's development of self-regulation, which underlies school readiness, early school literacy academic achievement, and positive peer relations.

DETAILED DESCRIPTION:
Aims of the current project are:

1. Refine the intervention model to address the child's adaptation to school and development of self-regulatory skills and underlying multiple dimensions of school success.
2. Examine and test the consistency of developmental models of problem behavior, emotional adjustment, and normative self-regulation in childhood.
3. Evaluate the long-term impact of intervention on risk pathways to later drug abuse and health-risking behaviors by examining early risk markers, including children's problem behavior, poor emotional adjustment, and lack of school readiness.

ELIGIBILITY:
Original Inclusion Criteria:

* Parents with children between ages two and three
* Currently enrolled with Women, Infants, and Children (WIC)
* To qualify for the original study, families needed to meet criteria for child, family, and sociodemographic risk. Specifically, families either had to meet "child risk" factors or they had to have at least two of the three factors present to qualify for the study. To meet criterion for child risk, scores must be at least one SD above the normative average on the Eyberg Intensity of Problems factors, the Bates difficulty (i.e. negative emotionality) factor, or the conflict factor of the Adult-Child Relationship Scale. Family risk was determined by a score of one SD above the normative average on maternal depressive symptoms or parenting daily hassles, having substance use/abuse problems, or teen parent status. Sociodemographic risk was established using educational attainment because all WIC participants met criteria for low income. Families in which educational attainment is less than three years of college for both parents satisfied the requirement of sociodemographic risk.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 731 (Actual)
Dates: Start 2003-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Home visit assessment | yearly
  Includes caregiver assessment packets (including CBCL, Eyberg, Rothbart Effortful Control scales, CESD-D, parental substance use, Adult-Child Relationship scale), child assessment (including DIBELS and Woodcock-Johnson) and Parent-Child videotaped interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Dishion, PhD, Principal Investigator — University of Oregon- Child and Family Center
Locations (3):
- United States (3):
  - University of Oregon-Child and Family Center, Eugene, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia